CLINICAL TRIAL: NCT01529372
Title: REnAL denervatIon by ultraSound Transcatheter Emission
Acronym: REALISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0020-HT
Record Dates: First submitted 2012-01-19; First posted 2012-02-08 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Resistant Hypertension
Keywords: Hypertension; Blood pressure; Renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous renal denervation (Experimental)
  Interventions: Device: PARADISE percutaneous renal denervation

INTERVENTIONS:
Device: PARADISE percutaneous renal denervation — Intravascular ultrasound emission
  Other Names: ReCor Medical PARADISE

SUMMARY:
The REALISE trial is a single-arm, open-label, prospective, post market evaluation to be conducted on twenty (20) eligible patients with a twelve month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension, as defined in the 2007 ESH-ESC guidelines
* 18 years of age or older
* Negative pregnancy test for female patients of childbearing potential
* Willing and able to comply with follow-up requirements
* Signed informed consent

Exclusion Criteria:

* Secondary hypertension
* Main renal arteries length < 20 mm
* Main renal arteries diameter < 4 mm
* Renal artery stenosis
* Iliac/femoral artery stenosis precluding insertion of the catheter
* Allergy to contrast media
* Currently participating in the study of an investigational drug or device
* Hemodynamics abnormality
* Moderate to severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of successful interventions | Up to 24 hours
  A successful intervention is defined by the ability to successfully:
  1. Introduce the PRDS catheter
  2. Position the PRDS catheter
  3. Deliver ultrasound energy
  4. Retrieve the PRDS catheter
Percentage of patients with device- or procedure-related adverse events | 12 months
  Anticipated adverse events include:
  * Puncture site-related events
  * Renal artery stenosis, aneurysm, dissection, or perforation
  * Renal infarction, acute kidney injury, or renal failure
  * Arterial and venous thromboembolic events (including myocardial infarction, stroke, aortic or peripheral artery disease, etc.)

SECONDARY OUTCOMES:
Change from baseline in ambulatory blood pressure | 12 months
Change from baseline in anti-hypertensive medication intake | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Montalescot, Professor, Principal Investigator — Hôpital Pitié-Salpêtrière
Locations (2):
- France (2):
  - Université de Toulouse et CHU, Toulouse
  - Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region